CLINICAL TRIAL: NCT06213493
Title: Role of the BACE1-AS Long Noncoding RNA in Ischemic Heart Failure
Brief Title: Bace1as Role in Heart Failure (BACE1AS-HF)
Acronym: BACE1AS-HF
Status: Completed | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Collaborators: Istituti Clinici Scientifici Maugeri di Pavia (Unknown)
Responsible Party: Principal Investigator, Fabio Martelli, Director of Molecular Cardiology Laboratory, IRCCS Policlinico S. Donato
Other Study IDs: BACE1AS_HF- RF-2019-12368521
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure; Acute Coronary Syndrome
Keywords: long noncoding RNA; heart failure; acute coronary syndrome; biomarkers
MeSH Terms: conditions — Heart Failure; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — blood, tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Non end-stage heart failure: Measurement of tissutal RNAs in non end-stage heart failure patients undergoing to left ventricle reconstruction
  Interventions: Diagnostic Test: measurement of RNAs
- ACS patients: Measurement of circulating RNAs in acute coronary syndrome (ACS) patients treated with percutaneous angioplasty and undergoing to ventricle remodelling
  Interventions: Diagnostic Test: measurement of RNAs
- HF patients: Measurement of circulating RNAs in heart failure patients
  Interventions: Diagnostic Test: measurement of RNAs
- Controls: Measurement of RNAs in individuals not affected by cardiovascular diseases
  Interventions: Diagnostic Test: measurement of RNAs

INTERVENTIONS:
Diagnostic Test: measurement of RNAs — RNAs will be measured in heart tissues and in peripheral blood mononuclear cells

SUMMARY:
The objective of this project is 1) to explore the clinical relevance of BACE1-AS and BACE1 as therapeutic targets and 2) to evaluate their potentiality as biomarkers in ischemic heart failure (HF).

The first aim will be studied by validating in left ventricle biopsies in patients with post-ischemic heart failure the transcriptome and DNA methylation status data obtained in cell lines where the expression of BACE1-AS has been modulated.

The investigation of BACE1-AS and BACE1 as biomarkers will be obtained by using peripheral blood mononuclear cells (PBMCs) from patients with acute coronary syndrome (ACS) treated with percutaneous angioplasty (PCI) procedure and undergoing to left ventricular remodeling. Furthermore, PBMCs from patients with chronic ischemic HF recruited from the Istituti Clinici Scientifici Maugeri Pavia will be also used. From the data obtained from these patients and from non-decompensated subjects, the levels of BACE1-AS and BACE1 in the blood will be measured and correlated with each other and with β-amyloid levels (βA), as well as with clinically relevant parameters.

DETAILED DESCRIPTION:
1.1) Validation of transcriptomic data obtained in vitro: The transcriptome of the AC16 cardiomyocyte cell line in which the expression of BACE1-AS was induced by lentivirus vectors will be analyzed, thus identifying the transcripts specifically modulated by BACE1-AS. The data obtained in vitro will be validated by analyzing the RNAs extracted from 20 HF patients and 20 controls. These RNA samples are already available thanks to the RNA_HF_AS project "Study of the transcriptome in heart failure and aortic stenosis" (San Raffaele Hospital - Milan, Ethics Committee CE 85/int/2016).

1.2) Validation of epigenetic data: The effect of BACE1-AS on the state of DNA methylation will be studied in the AC16 cardiomyocyte cell line. In over-expressing BACE1-AS cells, DNA hypomethylation will be evaluated by MS-HRM and pyrosequencing studies of bisulfite-modified genomic DNA of 69 enhancer sequences identified by us as candidates in preliminary studies. The data thus obtained will be validated in 20 cardiac biopsies from patients with post-ischemic HF and in 20 controls. Left ventricular biopsies will be taken after obtaining informed consent from 20 patients suffering from non-terminal dilated cardiomyopathy (DCM) undergoing left ventricular reconstruction (SVR) surgery at the San Donato Policlinico. A sufficient number of samples with these characteristics have already been obtained from IRCCS Policlinico San Donato as part of the RNA_HF_AS project (San Raffaele Hospital - Milan, Ethics Committee CE 85/int/2016). and not completely used for the study.

1.3) Study of the expression levels of BACE1-AS, BACE1 in PBMC of patients with ischemic cardiomyopathy.

The expression levels of BACE1 and BACE1-AS will be measured in PBMCs from the following groups:

Group 1:

130 ACS patients with left ventricular systolic dysfunction (left ventricular ejection fraction (LVEF) < 45%) at 12 months follow-up after PCI, as well as 100 control subjects, recruited from the Interventional Cardiology Unit of the IRCCS Policlinico San Donato. The measurements of BACE1, BACE1-AS and βA will be carried out at the Molecular Cardiology Laboratory of the IRCCS Policlinico San Donato. These activities are included among those approved in the RNA_ACS protocol (Ethics Committee of the San Raffaele Hospital - Milan 14/int/2020) "RNA as prognostic biomarkers in patients with acute coronary syndrome"

Group 2:

240 patients with chronic post-ischemic HF and 120 age/sex-matched healthy controls. The recruitment of this group and measurements of BACE1, BACE1-AS and βA will be carried out at the Istituti Clinici Scientifici Maugeri Pavia.

ELIGIBILITY:
1. Left ventricular biopsies from patients with post-ischemic HF

   Inclusion Criteria:
   * left ventricular reconstruction surgery (SVR)
   * ESVI >35 ml/m2
   * EF<40%
   * previous anterior transmural infarction
   * age 40-75 years

   Exclusion Criteria:
   * ESVI <35 ml/m2
   * EF>40%
   * Tempo from E unknown
   * Pregnant women
   * Patients with genetic diseases
   * Patients suffering from malignant neoplasm
   * Subjects with collagenopathies
   * Subjects undergoing chemo/radiotherapy
   * Subjects undergoing prolonged steroid therapy
   * Subjects with known active infectious diseases
   * Subjects with positive serology for HIV, HBV (not vaccinated), HCV.
2. Patients with ACS and left ventricular dysfunction 12 months after percutaneous angioplasty

   Inclusion criteria:
   * Age >18 years
   * Patients with ACS (first episode), defined according to the ESC 2017 guidelines [19]
   * Informed consent to enrollment in the study

   Exclusion Criteria:
   * Severe heart valve disease or other conditions requiring cardiac surgery
   * Previous cardiac surgery including coronary artery bypass grafting
   * Total chronic occlusions
   * Patients with known hypersensitivity or contraindication to any of the following drugs:

   heparin aspirin, clopidogrel, ticlopidine, sirolimus, everolimus.
   * Any contraindication to implantation of drug-eluting stents (DES)
   * Patients with previous documented myocardial infarction;
   * LVEF <30% before PCI
   * Patients in cardiogenic shock
   * Patients with advanced STEMI (> 48 h from the onset of symptoms/Q waves on ECG) or undergoing fibrinolysis;
   * Patients with known previous cardiomyopathy with LVEF < 40%
   * Patients suffering from malignant neoplasms or systemic pathologies with a quoad vitam prognosis of less than 1 year;
   * Patients suffering from known active infectious diseases;
   * Patients who are unable to express valid informed consent at the time of enrollment
   * Pregnant women
3. Patients with chronic post-ischemic HF ( recruitment at the Istituti Clinici Scientifici Maugeri Pavia)

Inclusion criteria:

1. All patients admitted to Rehabilitation Cardiology at the Cardiology Department of ICS Maugeri with a diagnosis of chronic heart failure on an ischemic or "acute" basis due to exacerbation of chronic heart failure due to previous ischemia and whose therapies have been optimized at the moment of enlistment.
2. NYHA Class II-III at the time of enlistment;
3. Age over 18 years;
4. Informed consent signed at the time of enrollment in the study.

Exclusion criteria:

1. Denial of informed consent;
2. End-stage renal disease;
3. Presence of ACS, stroke, transient ischemic attack, major cardiovascular surgery, percutaneous coronary angioplasty or carotid angioplasty in the previous 3 months;
4. Patients undergoing cardiac transplantation or on the active list for cardiac transplantation or undergoing LVAD implantation;
5. Presence of hemodynamically significant mitral or aortic valve disease except mitral insufficiency due to ventricular dilatation;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Left ventricular biopsies from patients with post-ischemic HF. Left ventricular tissue fragments from patients with post-ischemic HF undergoing to left ventricular reconstruction (SVR) will be used
  2. Patients with acute coronary syndrome and left ventricular dysfunction 12 months after percutaneous angioplasty Control group will be represented by patients suffering from unstable angina.
  3. Patients with chronic post-ischemic HF (recruitment at the Istituti Clinici Scientifici Maugeri Pavia ICS) All patients admitted with a diagnosis of chronic heart failure or an ischemic or "acute" basis due to exacerbation.
Sampling Method: Probability Sample
Enrollment: 630 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Cardiac tissutal RNAs expression | From year 1 to year 3
  The RNAs cardiac tissutal expression of non- and end-stage heart failure patients compared to controls
Peripheral blood RNAs expression in ACS | From year 1 to year 3
  The RNAs expression in peripheral blood mononuclear cells of acute coronary syndrome patients treated with percutaneous angioplasty and remodelling compared to controls
Peripheral blood RNAs expression in heart failure | From year 1 to year 3
  The RNAs expression in peripheral blood mononuclear cells of heart failure patients compared to controls

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Martelli, PhD, Principal Investigator — IRCCS Policlinico S. Donato
Locations (1):
- Irccs Policlinico San Donato, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: No